CLINICAL TRIAL: NCT07293039
Title: Effects of Isometric Gluteal Activation Plus Movement Retraining vs. Gluteal Activation Alone on the Forward Step-Down Test
Brief Title: Gluteal Activation Plus Movement Retraining
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003174
Record Dates: First submitted 2025-12-02; First posted 2025-12-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-11

CONDITIONS: Movement, Abnormal; Lower Extremity Problem
MeSH Terms: conditions — Dyskinesias

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator performing the data analysis will be blinded from the group allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluteal Activation Group (Active Comparator): The Control group will receive an HEP focusing on isometric gluteal activation.
  Interventions: Other: Control HEP focusing on isometric gluteal activation
- Gluteal Activation Plus Movement Training Group (Experimental): The Experimental group will receive an HEP focusing on isometric gluteal activation plus movement retraining program.
  Interventions: Other: Experimental HEP focusing on isometric gluteal activation plus a movement retaining program

INTERVENTIONS:
Other: Control HEP focusing on isometric gluteal activation — All participants will receive the HEP for hip muscle activation training. The HEP for hip musculature activation consists of five isolated hip activation exercises including side-lying clams, side-lying clams with trunk activation via side-plank, side-lying hip abduction, side-lying hip abduction with trunk activation via side-plank, and fire hydrants all of which improve hip gluteal recruitment.
  After the 4th week, both groups are to return to the clinic and asked to briefly perform exercises from their HEP so that their form can be reassessed with any modifications if needed along with any questions that they may have. Each participant following the 8-week period will be scheduled to return to the clinic to turn in their compliance form and perform follow-up surface electromyography (sEMG), weight, and FSDT using the same procedures as before.
  Arms: Gluteal Activation Group
Other: Experimental HEP focusing on isometric gluteal activation plus a movement retaining program — Only participants in the experimental group will receive the movement retraining program HEP. The HEP will be a combination of single leg Romanian Deadlift (RDL), single leg squat, and standing split squat that have been used in previous research and are proved to get significant gluteus medius (Gmed) activation. They will also participate in the gluteal activation HEP program that have been proved to increase hip musculature recruitment, as performed by the control group.
  After the 4th week, both groups are to return to the clinic and asked to briefly perform exercises from their HEP so that their form can be reassessed with any modifications if needed along with any questions that they may have. Each participant following the 8-week period will be scheduled to return to the clinic to turn in their compliance form and perform follow-ups sEMG, weight, and FSDT using the same procedures as before.
  Arms: Gluteal Activation Plus Movement Training Group

SUMMARY:
The purpose of this study is to determine if an isometric gluteal activation home exercise program (HEP) combined with a movement retraining program utilizing feedback cues produces significant changes in scores on the Forward Step-Down Test (FSDT) in healthy young adults with movement coordination impairments.

Aim 1: To determine if an isometric gluteal activation HEP with a movement retraining program with feedback cues produces significant changes on scores FSDT compared to the gluteal activation HEP alone.

Aim 2: To determine if an isometric gluteal activation HEP followed with a movement retraining program with feedback cues produces significant changes on category FSDT compared to gluteal activation HEP alone.

Aim 3: To determine if an isometric gluteal activation HEP with a movement retraining program with feedback cues produces changes in the peak activation of the gluteus medius (GMed) and gluteus maximus (GMax) during the FSDT compared to the gluteal activation HEP alone.

Aim 4: To determine if an isometric gluteal activation HEP with a movement retraining program with feedback cues produces changes in the mean activation of the GMed and GMax during the FSDT compared to the gluteal activation HEP alone.

Aim 5: To determine if HEP dose has an effect on the FSDT response, as measured by change in score on the FSDT.

ELIGIBILITY:
Inclusion Criteria:

* Participants must between the ages of 18 and older, if they were healthy via the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+), and scored a 2 or higher on the FSDT.

Exclusion Criteria:

* Participants have any current knee/hip pain, past knee/hip pathology in the past 3 months on their dominant leg or that the participant believes would impact their ability to participate in the study, or any past lower extremity (LE) surgery in their dominant leg that the participant believes would impact their ability to participate in the study, a concussion in the past 3 months, or if they have any vestibular pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2026-01-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Forward Step-Down Test (FSDT) | Baseline and after 8-week Home Exercise Program (HEP) intervention.
  Rating on the FSDT (0-6; 0-1 = good movement quality, 2-3 = moderate movement quality, 4 or more = poor movement quality).

SECONDARY OUTCOMES:
Peak Maximal Volitional Isometric Contraction (MVIC) on Gluteus Maximus (GMax). | Baseline and after 8-week HEP intervention.
  Peak activation (percent of maximal volitional isometric contraction [%MVIC]) of GMax during performance of the FSDT
Peak Maximal Volitional Isometric Contraction (MVIC) on Gluteus Medius (GMed). | Baseline and after 8-week HEP intervention.
  Peak activation (%MVIC) of GMed during performance of the FSDT
Mean Maximal Volitional Isometric Contraction (MVIC) on Gluteus Maximus (GMax). | Baseline and after 8-week HEP intervention.
  Mean activation (% MVIC) of GMax during performance of the FSDT
Mean Maximal Volitional Isometric Contraction (MVIC) on Gluteus Medius (GMed). | Baseline and after 8-week HEP intervention.
  Mean activation (% MVIC) of GMed during performance of the FSDT
HEP Compliance - Dose Response Relationship with FSDT and MVIC outcomes | After 8-week intervention.
  Self-reported completion of each HEP session will be recorded by the participant and then returned to the investigators post-completion

CONTACTS AND LOCATIONS:
Overall Officials: Erin McCallister, PT, DPT, Principal Investigator — LSU Health Sciences Center at Shreveport
Locations (1):
- LSU Health Sciences Center at Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powers CM. The influence of abnormal hip mechanics on knee injury: a biomechanical perspective. J Orthop Sports Phys Ther. 2010 Feb;40(2):42-51. doi: 10.2519/jospt.2010.3337. PMID 20118526
- [Background] Nascimento MB, Vilarinho LG, Lobato DFM, Dionisio VC. Role of gluteus maximus and medius activation in the lower limb biomechanical control during functional single-leg Tasks: A systematic review. Knee. 2023 Aug;43:163-175. doi: 10.1016/j.knee.2023.05.005. Epub 2023 Jul 7. PMID 37422984
- [Background] Wilczynski B, Zorena K, Slezak D. Dynamic Knee Valgus in Single-Leg Movement Tasks. Potentially Modifiable Factors and Exercise Training Options. A Literature Review. Int J Environ Res Public Health. 2020 Nov 6;17(21):8208. doi: 10.3390/ijerph17218208. PMID 33172101
- [Background] Branco GR, Resende RA, Bittencourt NFN, Mendonca LD. Interaction of hip and foot factors associated with anterior knee pain in mountain bikers. Phys Ther Sport. 2022 May;55:139-145. doi: 10.1016/j.ptsp.2022.04.001. Epub 2022 Apr 5. PMID 35413665
- [Background] McCallister E, Hughs C, Smith M, Flowers DW. Does a Hip Muscle Activation Home Exercise Program Change Movement Patterns on the Forward Step-Down Test? J Sport Rehabil. 2024 Jul 12;33(6):452-460. doi: 10.1123/jsr.2023-0372. Print 2024 Aug 1. PMID 38996451
- [Background] McCallister E, Bonvillain A, Christy A, Sensley C, & Flowers, DW. Effect of Adding Single-Leg Balance Training With a Hip Muscle Activation Program on Frontal Plane Movement Quality: A Randomized Controlled Trial in Adult Females. Women Sport Phys Act J. 2025;33(1):1-16. doi:10.1123/wspaj.2024-0091
- [Background] Peleg S, Pelleg-Kallevag R, Almog Y, Herman G, Nakdimon O, Arnon M, Dar G. Forward step down test - clinical rating is correlated with joint angles of the pelvis and hip: an observational study. BMC Musculoskelet Disord. 2023 Oct 12;24(1):807. doi: 10.1186/s12891-023-06943-4. PMID 37828484
- [Background] Davis IS, Tenforde AS, Neal BS, Roper JL, Willy RW. Gait Retraining as an Intervention for Patellofemoral Pain. Curr Rev Musculoskelet Med. 2020 Feb;13(1):103-114. doi: 10.1007/s12178-020-09605-3. PMID 32170556
- [Background] Chua LK, Jimenez-Diaz J, Lewthwaite R, Kim T, Wulf G. Superiority of external attentional focus for motor performance and learning: Systematic reviews and meta-analyses. Psychol Bull. 2021 Jun;147(6):618-645. doi: 10.1037/bul0000335. PMID 34843301
- [Background] Moinuddin A, Goel A, Sethi Y. The Role of Augmented Feedback on Motor Learning: A Systematic Review. Cureus. 2021 Nov 18;13(11):e19695. doi: 10.7759/cureus.19695. eCollection 2021 Nov. PMID 34976475
- [Background] Collings TJ, Bourne MN, Barrett RS, Meinders E, GONcALVES BAM, Shield AJ, Diamond LE. Gluteal Muscle Forces during Hip-Focused Injury Prevention and Rehabilitation Exercises. Med Sci Sports Exerc. 2023 Apr 1;55(4):650-660. doi: 10.1249/MSS.0000000000003091. PMID 36918403
- [Background] Boren K, Conrey C, Le Coguic J, Paprocki L, Voight M, Robinson TK. Electromyographic analysis of gluteus medius and gluteus maximus during rehabilitation exercises. Int J Sports Phys Ther. 2011 Sep;6(3):206-23. PMID 22034614
- [Background] Distefano LJ, Blackburn JT, Marshall SW, Padua DA. Gluteal muscle activation during common therapeutic exercises. J Orthop Sports Phys Ther. 2009 Jul;39(7):532-40. doi: 10.2519/jospt.2009.2796. PMID 19574661
- [Background] Aiken CA, Fairbrother JT, Post PG. The effects of self-controlled video feedback on the learning of the basketball set shot. Front Psychol. 2012 Sep 11;3:338. doi: 10.3389/fpsyg.2012.00338. eCollection 2012. PMID 22973257
- [Background] van Melick N, Meddeler BM, Hoogeboom TJ, Nijhuis-van der Sanden MWG, van Cingel REH. How to determine leg dominance: The agreement between self-reported and observed performance in healthy adults. PLoS One. 2017 Dec 29;12(12):e0189876. doi: 10.1371/journal.pone.0189876. eCollection 2017. PMID 29287067
- [Background] Konrad P. The ABC of EMG: A Practical Introduction to Kinesiological Electromyography. Noraxon U.S.A.; 2006.
- [Background] Harput G, Ulusoy B, Akmese R, Ergun N. Comparison of muscle activation levels and knee valgus between individuals with medial patellofemoral ligament reconstruction and healthy individuals during fatiguing step down task. Clin Biomech (Bristol). 2020 Aug;78:105067. doi: 10.1016/j.clinbiomech.2020.105067. Epub 2020 Jun 6. PMID 32535475
- [Background] Selkowitz DM, Beneck GJ, Powers CM. Which exercises target the gluteal muscles while minimizing activation of the tensor fascia lata? Electromyographic assessment using fine-wire electrodes. J Orthop Sports Phys Ther. 2013 Feb;43(2):54-64. doi: 10.2519/jospt.2013.4116. Epub 2012 Nov 16. PMID 23160432
- [Background] Selkowitz DM, Beneck GJ, Powers CM. Comparison of Electromyographic Activity of the Superior and Inferior Portions of the Gluteus Maximus Muscle During Common Therapeutic Exercises. J Orthop Sports Phys Ther. 2016 Sep;46(9):794-9. doi: 10.2519/jospt.2016.6493. Epub 2016 Aug 5. PMID 27494053
- [Background] Hopper AJ, Haff EE, Joyce C, Lloyd RS, Haff GG. Neuromuscular Training Improves Lower Extremity Biomechanics Associated with Knee Injury during Landing in 11-13 Year Old Female Netball Athletes: A Randomized Control Study. Front Physiol. 2017 Nov 7;8:883. doi: 10.3389/fphys.2017.00883. eCollection 2017. PMID 29163219
- [Background] Loudon JK, Wiesner D, Goist-Foley HL, Asjes C, Loudon KL. Intrarater Reliability of Functional Performance Tests for Subjects With Patellofemoral Pain Syndrome. J Athl Train. 2002 Sep;37(3):256-261. PMID 12937582

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT07293039/Prot_SAP_000.pdf